CLINICAL TRIAL: NCT04859543
Title: Prospective, Interventional Diagnostic, Multicenter, Non-treatment Clinical Study Identifying Specific Molecular Changes by Using Genomic Sequencing Technologies in Refractory/Recurrent or Very High-risk Pediatric CNS Tumors.
Brief Title: Pediatric Prospective Personalized Immune and Target Identification Trial
Acronym: PPROSPERITIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Masaryk University (Other)
Collaborators: Brno University Hospital (Other); Roche s.r.o. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KDO-2019-001
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Central Nervous System Neoplasms; Pediatric Cancer; GEN1 Gene Mutation; Tumor, Brain
Keywords: Pediatric oncology, CNS tumors, Personalized medicine
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic group (Other): Tumor and blood samples will be collected from each patient and broad molecular profiling will be performed. The results of the evaluation of the tumor specimens will determine if the patient's tumor has an actionable mutation for which treatment is available.
  Interventions: Device: FoundationOneHeme

INTERVENTIONS:
Device: FoundationOneHeme — Tumor tissue obtained during standard surgery will be subsequently examined histopathologically and the content of cancer cells will be determined. Broad molecular profiling of the tumor; with potential results finding such molecular changes, for which the specific targeted anti-tumor treatment will be performed.

SUMMARY:
PPROSPERITIT is a prospective clinical study assessing the use of comprehensive molecular profiling to define the best matching targeted and immune treatment for relapsed, refractory or very high risk pediatric CNS tumors.

DETAILED DESCRIPTION:
PPROSPERITIT will identify specific molecular changes by using genomic sequencing technologies in refractory/recurrent or very high-risk pediatric CNS tumors. The study will employ an analytically validated comparison of a selection of targeted agents/immune therapies on the basis of commercially available comprehensive genomic profiling FoundationOneHeme panel (F1Heme, comprising DNA and RNA analysis) vs selection of agents based on more complex DNA/RNA/Protein based analyses. This will be coupled to a computer algorithm that uses preexisting definitions and prioritization of target-agent pairs to assign patients by actionable mutation results to a targeted treatment. The selection of targeted agents will be performed by a multidisciplinary molecular tumor board, but the recommended treatment will not be a part of the PPROSPERTIT study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient Informed consent form must be appropriately obtained under the applicable local and regulatory requirements. Each patient must sign a consent form prior the enrollment to document their willingness to participate.
2. The subject is male or female, aged 1 - 19 years
3. The subject must have a histologically proven recurrent/ refractory or very high-risk CNS tumors
4. Patients must be in good overall physical condition, which allows tumor biopsy
5. Patients must have a life expectancy of at least 3 months.
6. Patients must have a tumor amenable to image-guided or direct vision biopsy and be willing and able to undergo a tumor biopsy and/or blood taking for molecular profiling.
7. Patients must be accessible for follow-up.

Exclusion Criteria:

1. Patients with known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
2. Pregnant and/or breastfeeding women, if applicable
3. No intention to treat the patient.

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients in which F1Heme molecular testing identified at least 1 clinically relevant alteration at the time of MTB decision. | Diagnostic assessment is done within 28 days from enrolment patient in the study.
  Evaluation of the feasibility of FoundationOneHeme

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslav Sterba, Prof, MD, Principal Investigator — University Hospital Brno
Locations (2):
- Czechia (2):
  - University Hospital Brno, Brno
  - Motol University Hospital, Prague

IPD SHARING:
Plan to Share IPD: No